CLINICAL TRIAL: NCT06918990
Title: Targeting the B Cell Response to Treat Antibody-Mediated Rejection With Carfilzomib and Belatacept (CarBel)
Brief Title: Treatment of Antibody-Mediated Rejection (ABMR) With CarBel
Acronym: CarBel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-42
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant Rejection
Keywords: Carfilzomib; Kidney transplant; Belatacept
MeSH Terms: interventions — carfilzomib; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Treatment Arm (Experimental): Study Entry to Month-3 participants will receive:
  * Steroid pulse/taper
  * Kyprolis® (Carfilzomib)
  * Nulojix® (Belatacept)
  * Tacrolimus
  * Mycophenolate
  * Prednisone
  After 3 months participants will receive:
  * Belatacept +
  * Mycophenolate
  * Prednisone
  * Tacrolimus
  Interventions: Biological: Carfilzomib; Biological: Belatacept
- Conventional Treatment Arm (Experimental): Study Entry to Month-3 participants will receive:
  * Steroid pulse/taper
  * Intravenous Immunoglobulin (IVIG)
  * Tacrolimus OR Belatacept +
  * Mycophenolate
  * Prednisone
  After 3 months participants will receive:
  * Kyprolis® (Carfilzomib)
  * Nulojix ® (Belatacept)
  * Tacrolimus
  * Mycophenolate
  * Prednisone
  After an additional 3 months (6 months from study entry) participants will receive:
  * Belatacept +
  * Mycophenolate
  * Prednisone
  * Tacrolimus
  Interventions: Biological: Carfilzomib; Biological: Belatacept

INTERVENTIONS:
Biological: Carfilzomib — Administered by intravenous infusion over 60 minutes.
  Other Names: Kyprolis
Biological: Belatacept — Administered by intravenous infusion over 30 minutes.
  Other Names: Nulojix

SUMMARY:
The purpose of this study is to see:

1. If using these two drugs (carfilzomib and belatacept) together is safe
2. If the use of these two study drugs in addition to the usual immunosuppression for kidney transplant patients can improve your transplanted kidney function by lowering the antibodies you have against your transplanted kidney
3. If the study drugs effect the immune cells that were responding to your donor kidney. And, whether blood or urine tests can measure signs of inflammation and kidney cell injury
4. If using new computer techniques can help describe important changes seen on biopsy in your donated kidneys

The primary objective is to assess the efficacy of carfilzomib and belatacept therapy when added to current treatment with steroids and maintenance immunosuppression, compared to conventional treatment alone, to improve the clinical outcome of renal transplant patients with active and chronic - active ABMR occurring more than 6 months after renal transplantation or less than 6 months post-transplant with persistent refractory Antibody-Mediated Rejection (ABMR)

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and agree to participate in the study.
2. Have received a kidney transplant from a living or deceased donor (including re-transplants).
3. Men and women must agree to use birth control during the study and for 3 months after the last dose of study drugs, or be surgically sterile or post-menopausal.
4. Heart function must be good enough (LVEF of at least 40%) without severe heart issues or high blood pressure in the lungs.
5. Must have been previously exposed to the Epstein-Barr Virus (EBV).
6. Diagnosed with specific types of kidney transplant rejection based on criteria, with certain conditions on timing and treatment history.
7. Kidney function must be at a certain level (eGFR of at least 30 ml/min/1.73 m²).
8. Specific scores related to kidney biopsy results must be within certain limits.
9. Must have a measurable level of specific antibodies against the donor kidney (HLA DSA) with a certain intensity.
10. Up-to-date vaccinations according to guidelines for transplant patients.
11. Must have a negative tuberculosis (TB) test and chest x-ray before enrollment, no symptoms or known contact with TB, and not have recently traveled to or lived in areas with high TB rates. If previously infected with TB, must have completed treatment and have a recent negative chest x-ray.
12. If previously infected with COVID-19, must be fully recovered for at least 21 days before joining the study. No COVID-19 test required for those without symptoms.

Exclusion Criteria:

1. Unable or unwilling to give consent or follow study rules.
2. Kidney transplant with incompatible blood types.
3. Very high levels of protein in urine, indicating severe kidney issues.
4. Previously had a non-kidney organ or bone marrow transplant.
5. Any other medical issues that might increase risk, make following the study rules hard, or affect study results, as judged by the study doctor.
6. Heart attack within the last year, uncontrolled chest pain, or signs of a recent heart problem on an ECG.
7. Severe heart failure (Class 3 or higher).
8. Irregular heartbeats that can't be controlled with medication.
9. Used any experimental drug within the last 4 weeks or longer if the drug stays in the body longer.
10. Serious medical or mental health issues that could interfere with the study.
11. Cancer diagnosis or treatment within the past 2 years, except for certain skin cancers or cancers with a high cure rate.
12. Known allergy to Captisol® (used in the study drug).
13. Very low blood counts (hemoglobin, neutrophils, or platelets).
14. Positive for HIV, Hepatitis B, or Hepatitis C, unless Hepatitis C was successfully treated.
15. Severe infections needing treatment in the last 4 weeks.
16. Specific kidney infection (BK nephropathy) or high levels of BK virus.
17. Certain kidney biopsy results indicating other types of rejection or kidney diseases.
18. Treated for a specific viral infection (CMV) in the last 90 days or resistant to certain CMV treatments.
19. Received a live vaccine in the last 4 weeks.
20. Severe liver disease or abnormal liver tests.
21. Pregnant or breastfeeding women. Women who can become pregnant must have a negative pregnancy test or proof they are not pregnant.
22. Any other significant medical condition that could interfere with the study according to the doctor.
23. Received certain antibody treatments in the last 3 months.
24. Kidney rejection within 6 months post-transplant without standard care.
25. Confirmed severe protein levels in urine.
26. Underwent certain treatments outside study criteria.
27. History of multiple unprovoked blood clots.
28. Diagnosed with Atypical Hemolytic Uremic Syndrome (aHUS).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of reduction in Microvascular Inflammation (MVI) >=2 points | 3-months post randomization and 12-months post receipt of Investigational Therapy (IT)
Part A: Incidence of reduction in the immunodominant donor-specific antibody (DSA) Mean Fluorescent Intensity (MFI) by >= 50% | 3-months post randomization and 12-months post receipt of IT
Part B: The incidence of 20% improvement in estimated Glomerular Filtration Rate (eGFR) using the Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI 2021) slope | 3-months post randomization and 12-months post receipt IT

SECONDARY OUTCOMES:
Change in albuminuria | 3-months post randomization and 12-months post receipt of IT
Change in Banff lesion grading score (2022 criteria) | 3-months post randomization and 12-months post receipt of IT
Change in immunodominant donor-specific antibody (DSA) MFI | 3-months post randomization and 12-months post receipt of IT
Change in estimated Glomerular Filtration Rate (eGFR) (2022 criteria) | 3-months post randomization and 12-months post receipt of IT
Incidence of Antibody-Mediated Rejection (ABMR) | 3-months post randomization and 12-months post receipt of IT
Incidence of Acute Cellular Rejection (ACR) | 3-months post randomization and 12-months post receipt of IT
Incidence of mixed ABMR/ACR | 3-months post randomization and 12-months post receipt of IT
Change in iBox scores | 3-months post randomization and 12-months post receipt of IT
Number of days hospitalized for administration of protocol | From entry to week 52
Number of days hospitalized for any other reason | From entry to week 52
Incidence of bacterial, viral, and fungal infections | From entry to week 52
Incidence of de novo malignancy | From entry to week 52
Time to all cause composite allograft loss | 3-months post randomization and 12-months post receipt of IT
  Allograft loss is defined as return to dialysis (continually for at least 30 days), allograft nephrectomy, re-transplantation, or death.
Time to all cause composite death-censored allograft loss | 3-months post randomization and 12-months post receipt of IT
  Death-censored allograft loss is defined as return to dialysis (continually for at least 30 days), allograft nephrectomy, or re-transplantation.
Time to patient death | 3-months post randomization and 12-months post receipt of IT

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Knechtle, M.D., Principal Investigator — Duke University Medical Center: Transplantation; Scott Sanoff, MD, Ph.D., Study Chair — Duke University Medical Center: Transplantation
Locations (10):
- United States (10):
  - University of Alabama Medical Center, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait